CLINICAL TRIAL: NCT00179569
Title: Molecular Processes of the Relaxation Response in Older Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004P-000418; H75-CCH-123424; H75-CCH-119124
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2007-11-05 (Estimated); Status verified 2007-11

CONDITIONS: Stress

INTERVENTIONS:
Behavioral: Relaxation response — 8 weeks of relaxation response training

SUMMARY:
The purpose of this study is to examine the molecular (nitric oxide) and biochemical (epinephrine, norepinephrine, cortisol and ACTH) parameters that are associated with RR elicitation and which may counteract the effects of acute stress in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* 60-80 years of age
* healthy individuals
* willing and able to attend treatment sessions
* willing to learn how to do and practice the relaxation-response
* access to a working telephone
* read and write English

Exclusion Criteria:

* Major medical or psychiatric illness
* asthma or seasonal allergies (resulting in nitric oxide levels >60 ppb)
* smoking
* previous relaxation-response practice
* current use of the following medications:systemic corticosteroids, anti-convulsants/psychotics, immunosuppressants, cytotoxic therapy, anabolic steroids, antidepressants (other than SSRIs), dicyclomine, bile acid binding resins, or sympathomimetic medication

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-08; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
A primary goal of this study is to quantify the magnitude of relaxation response elicitation by comparing oxygen consumption during rest versus during elicitation of the relaxation response in a sample of healthy older adults. | 8 weeks

SECONDARY OUTCOMES:
A second area of interest is the relationship between exhaled levels of nitric oxide (NO) and oxygen consumption (VO2) during relaxation response elicitation. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery A Dusek, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- BIDMC, Boston, Massachusetts, United States